CLINICAL TRIAL: NCT02024295
Title: Efficacy and Safety of S-adenosyl-l-methionine in Treatment of Alcoholic Hepatitis With Cholestasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XMX-AH-001
Record Dates: First submitted 2013-12-19; First posted 2013-12-31 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis, Alcoholic
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ademethionine (Experimental): ademethionine 1000mg ivgtt qd for 2 weeks, then orally 1000mg bid for 4 weeks.
  Interventions: Drug: Ademethionine
- Polyene Phosphatidyl choline (Active Comparator): Polyene Phosphatidyl choline 10ml ivgtt qd for 2 weeks, then Polyene Phosphatidyl choline 456 mg tid orally for 4 weeks.
  Interventions: Drug: Polyene Phosphatidyl choline; Drug: Ademethionine

INTERVENTIONS:
Drug: Ademethionine — ademethionine 1000mg ivgtt qd for 2 weeks, then orally 1000mg bid for 4 weeks.
  Other Names: ademethionine for 6 weeks
  Arms: Ademethionine
Drug: Polyene Phosphatidyl choline — Polyene Phosphatidyl choline 10ml ivgtt qd for 2 weeks, then Polyene Phosphatidyl choline 456 mg tid orally for 4 weeks.
  Other Names: Polyene Phosphatidyl choline for 6 weeks
  Arms: Polyene Phosphatidyl choline
Drug: Ademethionine — after 6 weeks of core treatment stage, then ademethionine 1000mg bid or qd orally for 42 weeks
  Other Names: stage 2, ademethionine for 42 weeks.

SUMMARY:
To determine the efficacy and safety S-adenosyl-l-methionine in alcoholic hepatitis with cholestasis.

DETAILED DESCRIPTION:
randomize first time for core treatment stage for 6 weeks, then randomized second time for extend treatment for 42 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index range 19-30kg/m2
* Alcohol Drinking history more than 5 years, for male ≥ 40g/ day, for female ≥ 20g/ day;
* STB from 2 to 10X ULN;
* ALP>1.5X ULN or GGT>3X ULN

Exclusion Criteria: any one of below,

* active virus hepatitis, or anti-HIV(+)
* exclude other hepatic disease: non-alcoholic fatty liver, drug-induced liver injury, autoimmune hepatitis( AMA/ANA>1:100), Wilson disease, hemochromatosis or other hepatic disease; obstructive cholestasis
* other non-hepatic diseases caused jaundice
* primary hepatic carcinoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
response rate of serum total bilirubin | 6 weeks
  response rate means percentage of subjects whose serum total bilirubin values declined from baseline over 30%

SECONDARY OUTCOMES:
level of serum direct bilirubin | 6 weeks and 48 weeks
level of serum bile acids | 6 weeks and 48 weeks
level of glutamic pyruvic transaminase | 6 weeks and 48 weeks
level of glutamic oxaloacetic transaminase | 6 weeks and 48 weeks
level of alkaline phosphatase | 6 weeks and 48 weeks
level of gamma-glutamyl transpeptidase | 6 weeks and 48 weeks
level of hyaluronic acid | 6 weeks and 48 weeks

OTHER OUTCOMES:
Liver biopsy | 48 weeks
  Liver biopsy is not demanded

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cheng, Principal Investigator — Beijing Ditan Hospital affiliated ffiated to Capital Medical University
Locations (2):
- China (2):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Jun Cheng, Beijing, Beijing Municipality